CLINICAL TRIAL: NCT02660268
Title: Evaluation of the Implementation of a Clinical Pathway for Improving the Performance of Medical and Surgical Management of Hip Prosthesis Infections
Brief Title: Contribution of a Clinical Pathway for the Treatment of Hip Prosthesis Infections
Acronym: OSCAR-PH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC14.455
Record Dates: First submitted 2016-01-12; First posted 2016-01-21 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Hip Prosthesis Infection
Keywords: Clinical pathway; Infection; Hip; Prosthesis
MeSH Terms: conditions — Infections | interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical pathway (Experimental): Patients in the experimental group will be followed according to the clinical pathway
  Interventions: Other: Clinical Pathway
- Control (No Intervention): Patients in the control group will receive standard care

INTERVENTIONS:
Other: Clinical Pathway — Implementation of a Clinical Pathway for Medical and Surgical Management of Hip Prosthesis Infections
  Arms: Clinical pathway

SUMMARY:
The main objective is to determine the contribution of a clinical pathway to improve the effectiveness of medico-surgical management of hip prosthesis infections in terms of clinical cure. The hypothesis raised is that the implementation of a clinical pathway would improve the performance of the medical and surgical management of chronic infections of prosthetic hip.

DETAILED DESCRIPTION:
The incidence of surgical site infections following the orthopedic surgery is about 1%. The number of prosthesis infections is estimated between 2000 and 2500 new cases a year in France.

Multiple medical and surgical care strategies are possible depending on the acute or chronic presentation, early or delayed antibiotic therapy; antibiotic therapy alone or associated with joint lavage, or with a prosthesis change in one or in two stages; after a long or short period of time, with or without fitting spacer. The practices are very heterogeneous for chronic infections depending on the terrain on which infection occurs and modalities of antibiotic therapy remain controversial. The treatment failure rate at 1 year is estimated at 20%.

The hypothesis raised is that the implementation of a clinical pathway would improve the performance of the medical and surgical management of chronic infections of prosthetic hip.

Objectives: To determine the contribution of a clinical pathway to improve the effectiveness of medico-surgical management of hip prosthesis infections in terms of clinical cure.

The secondary objectives are: To evaluate medical and surgical practices in diagnosis and treatment of hip prosthesis infections; identify the success factors and therapeutic failure of medical and surgical supported hip prosthesis infections in terms of clinical cure; determining management of quality indicators.

Methods: The clinical path will be developed by a committee of experts from the national and international recommendations, a review of the literature focused on the prosthesis conservation strategies and audit practices at the University Hospital of Grenoble.

The clinical path will be evaluated by an interventional trial clustered with control group, randomized, stepped wedge (inclusion staggered in time in 4 X 3 months) with an evaluation at one year.

The study population will include all patients treated for hip prosthesis infection in hospitals participating in the Alps, in a period of 16 months.

The primary endpoint will be the clinical cure at one year, defined as the absence of clinical signs of infection, inflammatory syndrome (C-Reactive Protein <10 mg / L), and radiological signs of infection.

Analysis: The association between the primary endpoint and the introduction of a clinical path will be quantified by the odds ratio estimated using a logistic regression model with adjustment for baseline characteristics of patients and inclusion of non-independence of observations.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years of age. Having a first episode of hip prosthesis infection defined by an infectious disease physician on clinical , radiological and microbiological criteria according the clinical practice guidelines of the French-Language Infectious Diseases Society May 13, 2009
* Signed Informed Consent
* Supported in one of the participating center (hospitals of Arc Alpin)
* Covered by health insurance

Exclusion Criteria:

* Subject < 18 years of age
* Inability to read and understand the participant's Information
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Clinical cure at 1 year of initial medical management, defined by the absence of the clinical signs of infection, the inflammatory syndrome (C- Reactive Protein <10 mg / L) and the radiological signs of infection | 12 months
  Clinical cure

SECONDARY OUTCOMES:
Time duration between first clinical signs and diagnosis | 12 months
Time duration between diagnosis and therapeutic management | 12 months
Total duration of antibiotic therapy | 12 months
Conservation or removal of hip prosthesis | 12 months
Cumulative length of hospital stay | 12 months
Gap analysis between observed care and the clinical path | 12 months
Functional sequelae at one year | 12 months
Quality of life at one year | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia PAVESE, MD, Principal Investigator — University Hospital, Grenoble
Locations (7):
- France (7):
  - Annecy Hospital, Annecy
  - Chambéry Hospital, Chambéry
  - University Hospital of Grenoble, Grenoble
  - Groupe Hospitalier Mutualiste de Grenoble., Grenoble
  - Hospices Civils de Lyon, Lyon
  - Hôpital Nord-CHU Saint Etienne, Saint-Etienne
  - Voiron Hospital, Voiron